CLINICAL TRIAL: NCT01452672
Title: Resource-sparing Radiotherapy for Breast Cancer
Brief Title: Resource-sparing Post-mastectomy Radiotherapy in Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Atomic Energy Agency (Other Government)
Collaborators: International Network for Cancer Treatment and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3.30.25
Record Dates: First submitted 2011-10-10; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Radiotherapy; Post-mastectomy; Molecular characterization
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT to chest wall and S/C (Active Comparator): Irradiation of the chest-wall and supraclavicular fossa
  Interventions: Radiation: Irradiation of the chest-wall and supraclavicular fossa
- RT to chest wall (Experimental): Irradiation of the chest-wall alone
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — RT 40 Gy in 15 fractions
  Arms: RT to chest wall
Radiation: Irradiation of the chest-wall and supraclavicular fossa — RT 40Gy in 15 fractions
  Arms: RT to chest wall and S/C

SUMMARY:
This study compares two different field set-ups in patients with breast cancer following a breast resection (mastectomy). These two set-ups are as follows: arm a - radiotherapy to the chest-wall only, and arm b - radiotherapy to the chest-wall and the supraclavicular fossa.

Patients in both treatment arms will receive radiotherapy with a shortened fractionation schedule.

Study hypothesis: irradiation of the chest-wall only is not inferior to irradiation of the chest-wall and supraclavicular fossa in terms of loco-regional control, survival and treatment toxicity.

DETAILED DESCRIPTION:
Post-mastectomy radiotherapy (PMRT) substantially reduces the risk of loco- regional failure as shown in several studies and meta-analyses. Two large trials for pre-menopausal node-positive breast cancer patients treated with mastectomy and chemotherapy showed that PMRT not only reduced loco- regional failure rates but also improved disease-free and overall survival rates.

Although the benefit of PMRT is clear, the optimal volume of tissues to be covered by the radiotherapy fields is controversial. Since the chest wall is the most likely location of recurrence, there is uniform consensus that the chest wall should be irradiated. However, areas of controversy exist regarding irradiation of the regional lymph nodes (axillary, supraclavicular and internal mammary lymph nodes), optimal radiation dose, and dose-fractionation.

If equivalent results could be achieved by omitting irradiation of the supraclavicular region in patients receiving adjuvant systemic therapy, this will simplify and expedite treatment in this patient population. Furthermore, the use of a shortened fractionation schedule of 40 Gy in 15 fractions (2.67 Gy per fraction) over 3 weeks which has been used in the UK and Canada for post-mastectomy patients for several decades will shorten the duration of treatment by reducing the number of patient visits for radiotherapy and increase the number of patients who can be treated. Treatment will be more convenient for patients and a reduction in the number of treatments could result in savings for strained health care systems.

This is a randomized comparison of two different radiotherapy field set-ups for post-mastectomy treatment of locally advanced breast cancer. Patients who have undergone modified radical mastectomy including axillary lymph node dissection will be randomized to receive one of two radiotherapy treatment arms, A and B following the completion of adjuvant chemotherapy. The radiotherapy for treatment Arm A consists of irradiation of the chest wall only while Treatment Arm B includes irradiation of the chest wall and the ipsilateral supraclavicular field. Patients on both treatment arms will receive radiation with a shortened fractionation schedule. Patients will be evaluated for local control, regional control, survival and treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be older than 18 and less than 81 years of age
2. WHO (ECOG) Performance Status of 0-2
3. Histologically confirmed diagnosis of infiltrating ductal carcinoma of the breast, lobular carcinoma or mixed (ductal and lobular) type.

   Note: Tumor diagnosis will be performed at the participating center according to the center's routine procedures.
4. Patients must have had a modified radical mastectomy (MRM) in which 6 or more axillary nodes were removed.
5. All patients should receive adjuvant chemotherapy following MRM. The initiation of radiation therapy must allow for the full recovery of blood counts (WBC > 3.0 x 109/L, Granulocytes > 1.5 x109/L and platelets > 75 x 109/L).

   Note: MRM should have been performed at maximum 3 months prior to the start of adjuvant chemotherapy.

   Special Note: Patients who have not received adjuvant chemotherapy will be required to receive adjuvant chemotherapy as per Appendix 3 prior to study entry and initiation of radiotherapy must allow for the full recovery of blood counts (WBC > 3.0 x 109/L, Granulocytes > 1.5 x109/L and platelets > 75 x 109/L MRM should have been performed within 3 months prior to the start of adjuvant chemotherapy.
6. Patients must have received adjuvant chemotherapy according to one of the two regimens found in Appendix 3.
7. Negative surgical margins by histopathology at the time of MRM. Note: Negative surgical margins means that there are no cancer cells at the inked margin of resection or otherwise at the margins of the mastectomy specimen.
8. The following indicators in the histological samples must be known :

   1. Tumor size
   2. Tumor site (quadrant, central, axillary tail)
   3. Presence of extensive intraductal component (EIC)
   4. Estrogen and Progesterone Receptor Status and the method of staining and detection.
   5. HER2 Status (optional), if given, the method must be provided.
9. Patients with the following TNM stages, all being M0: pT1 N1, pT2 N1, pT3 N0, pT0 N2, pT1 N2, pT2 N2, T3 N1, pT3 N2 (see Appendix 4 for TNM Stage)
10. Histological grades 1 - 3 (as per WHO criteria)
11. Patients must consent to return for scheduled treatments and follow up.
12. Written informed consent document signed

Exclusion Criteria:

1. Pathological pN3 (metastasis in 10 or more lymph nodes, clinically apparent internal mammary metastasis, metastasis in the supraclavicular lymph nodes)
2. Stages IIIB, IIIC and IV (any T4, any N3 or M1)
3. Recurrence of breast cancer following MRM and/or adjuvant chemotherapy.
4. Concomitant primary cancer in the contralateral breast.
5. History of other malignancy except carcinoma in situ of the cervix or non-melanoma skin cancer
6. Pregnant or breast-feeding
7. Previous chemotherapy other than adjuvant chemotherapy for treatment of the present breast cancer
8. Other severe concomitant disease that could impact upon the ability to deliver treatment or increase the risk of toxicity (such as uncompensated congestive heart failure, unstable coronary heart disease, uncompensated chronic obstructive pulmonary disease, collagen vascular diseases including systemic lupus erythematosus, systemic sclerosis, dermatomyositis, and ataxia telangiectasia).
9. Contraindications to radiation therapy (such as previous irradiation of the breast or chest wall)
10. Severe psychiatric disorder that may interfere with the process of informed consent and/or treatment or follow-up compliance.

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Local control. | 4 years
  The presence/absence of recurrent disease in the surgical scar, ipsilateral chest wall, ipsilateral skin and soft tissue.
Regional control. | 4 years
  The presence/absence of recurrent disease in the axilla, ipsilateral supraclavicular/infraclavicular nodes and or ipsilateral skin/soft tissue in the regional areas.
Overall survival. | 4 years
Disease-free survival. | 4 years
Acute adverse events. | 4 years
  During treatment and up to 90 days following the completion of treatment.
Late adverse events. | 4 years
  More than 90 days after the completion of radiation therapy.

SECONDARY OUTCOMES:
Patients' demographics. | 4 years
Reproductive history. | 1 year
  Number of pregnancies, miscarriages. Menstrual History.
Family history. | 1 year
  Family history of breast cancer.
Characterization of molecular profile of breast cancer patients. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rosenblatt, MD, Study Chair — International Atomic Energy Agency
Locations (9):
- Instituto Naciolal de Oncologia y Radiobiologia (INOR), Havana, Cuba
- Egypt (2):
  - Cairo National Cancer Institute, Cairo, Fom El-Khalig
  - Alexandria Ayadi Almostakbal Oncology Cenre., Alexandria
- Korle Bu Teaching Hospital, Accra, Ghana
- Institut National d'Oncologie, Rabat, Morocco
- University of Ibadan College Hospital, Ibadan, Nigeria
- Institut of Radiotherapy and Nuclear Medicine (IRNUM), Peshawar, Pakistan
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Cerraphasa Medical Faculty, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Nielsen HM, Overgaard M, Grau C, Jensen AR, Overgaard J. Loco-regional recurrence after mastectomy in high-risk breast cancer--risk and prognosis. An analysis of patients from the DBCG 82 b&c randomization trials. Radiother Oncol. 2006 May;79(2):147-55. doi: 10.1016/j.radonc.2006.04.006. Epub 2006 Apr 27. PMID 16647152
- [Background] Adenipekun A, Campbell OB, Oyesegun AR, Elumelu TN. Radiotherapy in the management of early breast cancer in Ibadan: outcome of chest wall irradiation alone in clinically nodes free axilla. Afr J Med Med Sci. 2002 Dec;31(4):345-7. PMID 15027777
- [Background] Truong PT, Olivotto IA, Whelan TJ, Levine M; Steering Committee on Clinical Practice Guidelines for the Care and Treatment of Breast Cancer. Clinical practice guidelines for the care and treatment of breast cancer: 16. Locoregional post-mastectomy radiotherapy. CMAJ. 2004 Apr 13;170(8):1263-73. doi: 10.1503/cmaj.1031000. PMID 15078851
- [Background] Owen JR, Ashton A, Bliss JM, Homewood J, Harper C, Hanson J, Haviland J, Bentzen SM, Yarnold JR. Effect of radiotherapy fraction size on tumour control in patients with early-stage breast cancer after local tumour excision: long-term results of a randomised trial. Lancet Oncol. 2006 Jun;7(6):467-71. doi: 10.1016/S1470-2045(06)70699-4. PMID 16750496
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- See also: International Atomic Energy Agency — http://www.iaea.org